CLINICAL TRIAL: NCT04268342
Title: Gonorrhoea Resistance Assessment by Nucleic Acid Detection: A Program Evaluation
Brief Title: Gonorrhoea Resistance Assessment by Nucleic Acid Detection (GRANDII)
Acronym: GRANDII
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Queensland (Other)
Collaborators: Kirby Institute (Other Government); Monash University (Other); South Australian Health and Medical Research Institute (Other); University of Melbourne (Other); University of California, Los Angeles (Other); Griffith University (Other); Queensland Health (Other Government); St Vincent's Hospital, Sydney (Other); SpeeDx Pty Ltd (Industry); NSW Health Pathology (Unknown); University of Sydney (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 17/180
Record Dates: First submitted 2020-02-06; First posted 2020-02-13 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-10

CONDITIONS: Drug Resistance, Microbial; Antimicrobial Stewardship; Gonorrhea
MeSH Terms: conditions — Gonorrhea

STUDY DESIGN:
Intervention Model Description: A before-after study design will be used to evaluate the proportion of all cases treated with ceftriaxone at return visit within standard care and the new management program respectively. Cure rates within the standard care and the new management program will also be assessed which will help illustrate the impact of the new management program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (No Intervention): When clinical services are in the standard case phase of the study, all cases of gonorrhoea infection diagnosed at those services will be managed according to current standard of care management guidelines i.e. all cases of gonorrhoea infection will be treated with ceftriaxone by injection plus oral azithromycin tablets as first line therapy, regardless of whether the treatment is given at the initial clinic or the return clinic visit.
- Implementation (Active Comparator): When clinical services are assigned to the implementation phase, first line treatment for gonorrhoea infection for patients treated at their first clinic visit will remain the same as it is currently: ceftriaxone by injection plus oral azithromycin tablets. However, patients who are not treated presumptively will be treated at their return visit on the basis of the drug resistance test results. Patients with gonorrhoea infection that is shown to be susceptible to ciprofloxacin will be treated with oral ciprofloxacin therapy when they return for review at clinical services in the implementation phase. Patients with gonorrhoea infection that is not susceptible to ciprofloxacin or with an indeterminate ciprofloxacin result will be treated with ceftriaxone by injection.
  Interventions: Other: Resistance guided treatment for gonorrhoea infection

INTERVENTIONS:
Other: Resistance guided treatment for gonorrhoea infection — For cases of gonorrhoea infection treated at the return visit, a nucleic acid assay will be used to determine individual eligibility for ciprofloxacin treatment
  Arms: Implementation

SUMMARY:
Three sexual health clinical services across Australia and their associated pathology testing laboratories are implementing a new management program for gonorrhoea infection. The services are implementing the use of gonorrhoea drug resistance testing as part of routine clinical and laboratory practice, where drug resistance test results are provided to clinicians quickly to guide choice of antibiotic therapy. Clinicians will identify gonorrhoea infection that is ciprofloxacin susceptible so that it can be treated with ciprofloxacin therapy, rather than ceftriaxone.

DETAILED DESCRIPTION:
This study aims to demonstrate the feasibility of a new approach to antibiotic stewardship based on individually tailored antibiotic prescribing. Three sexual health clinical services in New South Wales Australia with high caseloads of gay and bisexual men will adopt a new management practice for gonorrhoea infection involving provision of tailored antibiotic therapy by clinicians at the time of gonorrhoea diagnosis and treatment, guided by the results of resistance testing. The services are implementing the use of gonorrhoea drug resistance testing as part of routine clinical and laboratory practice, where drug resistance test results are provided to clinicians quickly to guide choice of antibiotic therapy. This differs from existing practice where the prolonged turn-around times for drug resistance testing results mean clinicians must prescribe drug therapy without knowing these results. This can lead to increasing levels of drug resistance to ceftriaxone.

The drug resistance test used in the new program detects genetic material (nucleic acids). It was developed and validated in Australia and is as accurate as existing culture-based drug resistance testing but provides quicker results. Patients treated presumptively at their first clinic visit will be treated with standard of care ceftriaxone. However, for cases treated at the return visit, clinicians will identify gonorrhoea infection that is ciprofloxacin susceptible so that it can be treated with ciprofloxacin therapy, rather than ceftriaxone. This will preserve ceftriaxone for situations where it must be used as the only effective drug available. Established patient follow-up procedures at clinical services will confirm that treatment has been successful.

Quantitative data from the clinical and laboratory services in the study will be used to assess the proportion of all cases treated with ceftriaxone. The cure rate in gonorrhoea cases within the new management program versus standard care will also be assessed which will help illustrate the impact of the new management program.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with gonorrhoea infection at the return visit

Exclusion Criteria:

* Patients for whom ciprofloxacin is contraindicated

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1626 (Estimated)
Dates: Start 2022-04-26 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Change in ceftriaxone use | 12 months after implementation commences
  The proportion of gonorrhoea cases treated at the return visit with ceftriaxone

SECONDARY OUTCOMES:
Cure rate | At 12 months after implementation commences
  The proportion of gonorrhoea cases treated at the return visit with a negative test of cure within 2-4 weeks within the new management program versus standard care
Acceptability | 1-12 months after implementation commences
  The acceptability of the new management program to clinic and laboratory staff and stakeholders will be assessed through a qualitative research study design. Service staff and external stakeholders will be selected purposively to take part in semi-structured in-depth interviews at different stages of the study. Sampling will be informed by data saturation. All interviews will be audio-recorded and transcribed verbatim. Qualitative data will be analysed using a system of thematic 'open' and 'axial' coding. Findings will be descriptive.
Cost effectiveness | 12 months after implementation commences
  The cost effectiveness of the new management program compared to standard care from the health service perspective
Process evaluation | 12 months after implementation commences
  To document the processes involved in the implementation of the new management program

CONTACTS AND LOCATIONS:
Overall Officials: David Whiley, PhD, Principal Investigator — The University of Queensland
Locations (1):
- University of Queensland, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data available at this stage.